CLINICAL TRIAL: NCT02681679
Title: Topical 0.1% Bromfenac Sodium for Intraoperative Pupil Dilation Maintenance and Prostaglandin E2 Inhibition in Femtosecond Laser-assisted Cataract Surgery
Brief Title: Topical 0.1% Bromfenac Sodium and Prostaglandin E2 Inhibition in Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Principle investigator, Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH), Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCPMOH2016-China-1
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.1% bromfenac ophthalmic solution (Experimental): Patients received 0.1% bromfenac ophthalmic solution twice a day for 3 days before surgery.
  Interventions: Drug: 0.1% bromfenac ophthalmic solution; Procedure: femtosecond laser cataract surgery
- control physiological normal saline (Placebo Comparator): Patients received control physiological normal saline twice a day for 3 days before surgery.
  Interventions: Procedure: femtosecond laser cataract surgery

INTERVENTIONS:
Drug: 0.1% bromfenac ophthalmic solution
  Arms: 0.1% bromfenac ophthalmic solution
Procedure: femtosecond laser cataract surgery

SUMMARY:
Since a new generation of femtosecond lasers became available for cataract surgery in 2009, the use of this image-guided system has provided several benefits, including a reduction in phacoemulsification energy by prefragmentation of the crystalline lens, and the potential advantages of more precise corneal incisions and capsulotomy formation. However, as with any new surgical technique, femtosecond laser cataract surgery also has potential complications. Intraoperative miosis is one of the most common intraoperative complications of femtosecond laser-assisted cataract surgery, with a reported prevalence ranging from 9.5 to 32.0%.8 Significant pupillary constriction necessitates the removal of the anterior capsule flap, fragmented nucleus and remaining cortex, which is potentially associated with a higher rate of surgery-related complications.

DETAILED DESCRIPTION:
Since a new generation of femtosecond lasers became available for cataract surgery in 2009, the use of this image-guided system has provided several benefits, including a reduction in phacoemulsification energy by prefragmentation of the crystalline lens, and the potential advantages of more precise corneal incisions and capsulotomy formation. However, as with any new surgical technique, femtosecond laser cataract surgery also has potential complications. Intraoperative miosis is one of the most common intraoperative complications of femtosecond laser-assisted cataract surgery, with a reported prevalence ranging from 9.5 to 32.0%. Significant pupillary constriction necessitates the removal of the anterior capsule flap, fragmented nucleus and remaining cortex, which is potentially associated with a higher rate of surgery-related complications.

Intraoperative miosis may be due to the intraocular effects that occur after femtosecond laser pretreatment. The intraocular tissues may be exposed to laser emissions, and lens proteins can be released into the anterior chamber. Together, these events trigger the release of unwanted cytokines. In a previous study, intraocular prostaglandin concentrations were found to be increased immediately after femtosecond laser pretreatment. Prostaglandins, especially prostaglandin E2 (PGE2), are known to play a role in inflammation-induced miosis.

Preoperative topical treatment with NSAIDs inhibits the release of prostaglandins in response to surgically-induced miosis by suppressing cyclooxygenase, the enzyme that transforms arachidonic acid into prostaglandin precursors. The effectiveness of ophthalmic NSAIDs in preventing miosis has been well documented in conventional phacoemulsification cataract surgery. However, whether this effect is also applicable to femtosecond laser-assisted cataract surgery is unknown. Yeoh has suggested the addition of NSAID eye drops to the dilation regimen during femtosecond laser cataract surgery, but no randomized study has been conducted to support this theory. Given the increasing popularity of femtosecond laser-assisted cataract surgery, the investigators sought to study whether topical NSAIDs might be beneficial in pupil maintenance and PGE2 inhibition during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* if they were 50 years of age or older and were scheduled to undergo femtosecond laser cataract surgery

Exclusion Criteria:

* a previous history of intraocular surgery;
* recent trauma;
* uveitis;
* systemic disease, such as diabetes mellitus; hypertension;
* the use of systemic or topical NSAIDs within 1 week of enrollment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pupil area measured using ImageJ software A | surgery
PGE2 levels measured with an enzyme-linked immunoassay | 2 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D. Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Nagy Z, Takacs A, Filkorn T, Sarayba M. Initial clinical evaluation of an intraocular femtosecond laser in cataract surgery. J Refract Surg. 2009 Dec;25(12):1053-60. doi: 10.3928/1081597X-20091117-04. PMID 20000286
- See also: Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/